CLINICAL TRIAL: NCT02321774
Title: Validation of a Wearable Sensor for Stress Response in a Virtual Reality Environment
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Steven Steinhubl, Principal Investigator, Scripps Translational Science Institute
Other Study IDs: IRB-14-6485
Record Dates: First submitted 2014-12-09; First posted 2014-12-22 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Stress; Virtual Reality; Wearable Sensor; Wellness

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Monitor stress response in a virtual reality environment using a wearable sensor to analyze and track heart rate variability (HRV).

DETAILED DESCRIPTION:
Wearable sensor technology is being developed that may allow, for the first time, the ability for individuals to better recognized their level of stress in any given situation on a continuous basis. A major focus of many of these wearable sensors is being able to accurately analyze and track heart rate variability (HRV), which is indicative of primarily parasympathetic/vagal tone and emotional state.3 However there is a need to validate the reliability of this measured response and understand any inter-individual variability.

The present study will take advantage of virtual reality scenarios to expose healthy volunteers to controlled stressful situations during monitoring with several standardized lab-based non-invasive physiological sensors as well as a novel wrist band sensor device to track individual response to stress.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 18

Exclusion Criteria:

* History of seizures
* History of vertigo or other vestibular abnormalities
* History of a chronic anxiety disorder
* History of cardiovascular disease or heart disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be made up of 50 adult men and women who are in general good health. Individuals will be recruited locally through fliers, word of mouth and email blasts to the Scripps community.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Changes in heart rate variability (HRV) as detected by the wristband sensor relative to measures of stress noted by lab-based physiologic monitoring equipment. | ~Four hours
  Collect continuous physiological data in real-time from participants undergoing a set of standardized stress exposure experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Steinhubl, MD, Principal Investigator — STSI
Locations (1):
- Virtual Reality Medical Center, San Diego, California, United States